CLINICAL TRIAL: NCT02828202
Title: Constitution of a National Cohort of Patients With Metastatic Melanoma Resectable Stage II or Stage III or IV or Unresectable Primary With the Objective of Setting up Epidemiological Monitoring and Clinico-biological Database, MELBASE
Brief Title: Follow-up of a National Cohort of Melanoma Resectable Stage II, Stage III or IV Patients or Unresectable Primary
Acronym: MelBase
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID-RCB 2015-A00138-41; 2011-244 (Other Grant/Funding Number: National Cancer Institute (INCa))
Record Dates: First submitted 2015-10-20; First posted 2016-07-11 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Skin; Biobank
MeSH Terms: conditions — Melanoma | interventions — Biological Products; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Primary melanoma (mostly paraffin embedded), metastatic sample (s)(paraffin embedded and frozen) from at least 1 site at inclusion and during evolution (particularly before treatment modification if clinically required, DNA and RNA from peripheral blood mononuclear cells, plasma, serum, peripheral blood mononuclear cells sampled at inclusion, every 6 months and before each new systemic therapy during 3 years.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prospective cohort Resectable stage II or III: Patients with resectable stage II or III melanoma
  Interventions: Other: Biological; Other: Tissular; Other: Quality of life
- Prospective cohort Unresectable stage III or stage IV (resectable or not) or unresectable primary: Patients with unresectable stage III, or stage IV (resectable or not) or unresectable primary melanoma
  Interventions: Other: Biological; Other: Tissular; Other: Quality of life

INTERVENTIONS:
Other: Biological — DNA from peripheral blood mononuclear cells, RNA, plasma, serum sampled at inclusion, every 6 months and before each new systemic therapy.
Other: Tissular — Primary melanoma (mostly paraffin embedded), metastatic sample (s)(paraffin embedded and frozen) from at least 1 site at inclusion and during evolution, particularly before treatment modification if clinically required.
Other: Quality of life — Specific questionnaires (FACT-M, EUROQUOL) at inclusion, every 3 months and before each new systemic therapy.

SUMMARY:
Prevention of melanoma can be efficient but mortality remains unchanged and 15 to 20% of patients still die from melanoma. Indeed metastatic melanoma is a heterogeneous highly and multiple mutations driven cancer. Significant survival benefit was demonstrated since 2011 with anti-CTLA4 +/- programmed death-1 (anti PD1) antibodies, B-Raf proto-oncogene, serine/threonine kinase (BRAF) and MAP-ERK kinase (MEK) inhibitors. Future improvement of advanced melanoma prognosis will rely on clinico-epidemiological studies and on biological studies to validate and identify new prognostic and predictive factors based on clinico-epidemiological and histological data, genomic host and tumor alterations, tumor microenvironment characteristics, individual immunological profile and functional imaging. In the context of marketing of costly innovative molecules, prospective collection of economic data on treatment and toxicity are required. Large biobanks collecting data from cohorts of advanced melanoma are mandatory for such projects.

MELBASE is a French prospective national cohort enrolling advanced melanoma patients whose objectives are to :

* provide an annual instrument panel with descriptive and correlative analysis of advanced melanoma patients in France including epidemiological, clinical, biological and economic characteristics
* validate and identify new clinical, epidemiological, and biological prognostic factors such as genomic host and tumor alterations, tumor microenvironment characteristics, individual immunological profile in advanced melanoma
* evaluate the risk-benefit, quality of life, the management cost of patients treated with validated and future treatments. The project also aims to define predictive biomarkers of response and toxicity including pharmacogenetics and tumor genetics alterations, tumor microenvironment characteristics, individual immunological profile.

Patients with resectable stage II or III will be enrolled since June 2023 with a 10 years follow-up.

Patients with unresectable stage III or IV (resectable or not) or unresectable primary melanoma will be enrolled prospectively since March 2013 with a 10 years follow-up (up to 6000 patients) from 27 French centers.

DETAILED DESCRIPTION:
Melanoma is on of rare cancer with increasing frequency in France. Prevention can be efficient in detecting melanoma with good prognosis but mortality remains unchanged and 15 to 20% of patients still die from melanoma. Indeed metastatic melanoma is a heterogeneous highly and multiple mutations driven cancer which is highly resistant to conventional treatments. Significant survival benefit was demonstrated since 2011 with anti-CTLA4 +/- anti PD1 antibodies and BRAF and MEK inhibitors.

In 2019, melanoma treatment with anti-PD1 antibodies or BRAFi+MEKi (dabrafenib+trametinib) was approved in stage III patients. Since 2023, in France, pembrolizumab is also approved for stage IIB/IIC melanoma patients ; thus, adjuvant therapy will be generalized without any sentinel lymph node surgery.

In addition, patients could also be treated by neoadjuvant therapies (pembrolizumab or clinical trial) in case of macroscopique stage III, pauci-metastatic stage IV or in case of rare stage II without surgery.

Future improvement of advanced melanoma prognosis will rely on clinico-epidemiological or biological studies to validate and identify new prognostic and predictive factors, also based on upon clinico-epidemiological and histological data, genomic host and tumor alterations, tumor microenvironment characteristics, individual immunological profile and functional imaging. In the context of marketing of costly innovative molecules, an assessment of resource consumption is required, with prospective collection of economic data on treatment and toxicity. Large biobanks collecting data from cohorts of advanced melanoma are mandatory for such projects.

Thus, MELBASE is a French national clinical biobank whose objectives are to:

* provide an annual instrument panel with descriptive and correlative analysis of advanced melanoma patients in France including epidemiological, clinical, biological and economic characteristics
* validate and identify new clinical, epidemiological, and biological prognostic factors such as genomic host and tumor alterations, tumor microenvironment characteristics, individual immunological profile in advanced melanoma
* evaluate the risk-benefit, quality of life, the management cost of patients treated with validated and future treatments. If possible, cost-effectiveness ratios will be calculated either in all treated patients or in selected populations of patients (based on clinical or biological criteria, like biomarkers), in order to identify populations where these new therapeutics will be the most cost-effective.

The project also aims to define predictive biomarkers of response and toxicity including pharmacogenetics and tumor genetics alterations, tumor microenvironment characteristics, individual immunological profile.

Patients with resectable stage II or III will be enrolled since June 2023 with a 10 years follow-up.

Patients with unresectable stage III or IV (resectable or not) or unresectable primary melanoma will be enrolled prospectively since March 2013 with a 10 years follow-up (up to 6000 patients) from 27 French centers.

The information collected in MELBASE will include clinical constitutional factors, factors linked to primary melanoma, factors linked to previous lymph node involvement, tumor kinetics informations, "American Joint Committee on Cancer" (AJCC) stage at inclusion and after various therapeutic intervention, serological markers, metastatic tumor genotyping (one or more sites, one or more time points), therapeutic interventions (medical, surgical, radiotherapy and palliative strategies) with evaluation of response, tolerance, medical direct costs, impact on quality of life,informations on COVID-19 infection and vaccination, consequences on melanoma treatment, date of death, date of latest news.

A virtual Tumor bank collecting samples (optional) mentions available samples stored each participating centers' Biological Resource Centers (BRC) : primary melanoma (mostly paraffin embedded), metastatic sample (s)(paraffin embedded and frozen) from at least 1 site at inclusion and during evolution (particularly before treatment modification if clinically required), DNA from peripheral blood mononuclear cells, plasma/serum sampled at inclusion, every 6 months and at each new treatment line during 3 years.

All date will be collected and organized on a data warehouse to generate clinico-epidemiological reports, analysis and a virtual catalog of biological material.

MELBASE project is consistent with the ethical chart of the hospital tumor banks published by the national French Cancer Institute (INCa). MelBase will also be managed by a chart ensuring each participating center management autonomy and availability of collected data A multidisciplinary scientific advisory board will identify research priorities based on clinical practice and scientific knowledge.

ELIGIBILITY:
1. Cohort Patients with Resectable stage II or III

   Inclusion Criteria:

   Patients diagnosed with resectable stage IIA/IIB/IIC or III melanoma, confirmed by histological exam.

   Naïve of systemic treatment for resectable stage II or III. Whose metastatic tumoral material can be collected by the Biological Resource Centers (optional criteria).

   Aged ≥ 18 years. Consenting to participate (signed informed consent).

   Exclusion Criteria:

   Patients refusal. Choroid melanoma. Resectable stage 1 melanoma. Stage 4, unresectable primitive or unresectable stage 3 melanoma. Patients under guardianship and under trusteeship.
2. Cohort patients with Unresectable stage III or stage IV (resectable or not) or unresectable primary:

Inclusion Criteria:

Patients diagnosed with an advanced melanoma, confirmed by histological exam. Unresectable primitive or unresectable stage III or stage IV (resectable or not) melanoma ; or patients treated by neoadjuvant treatment (exceptional) Naïve of systemic treatment for unresectable primitive or unresectable stage III or stage IV (resectable or not) melanoma, except adjuvant treatment.

Whose metastatic tumoral material can be collected by the Biological Resource Centers (optional criteria).

Aged ≥ 18 years. Consenting to participate (signed informed consent).

Exclusion Criteria:

Resectable stage 1, 2 or 3 melanoma. Patients refusal. Choroid melanoma. Patients under guardianship and under trusteeship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Cohort Patients with Resectable stage II or III melanoma.
  2. Cohort Patients With Metastatic Melanoma Stage IV (resectable or not) or Unresectable Stage III or unresectable primary.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  With a Kaplan-Meier curve analysis and Cox model

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 10 years
  With a Kaplan-Meier curve analysis and Cox model
Overall response | 10 years
  Determined by tumor assessments
Nature and incidence of Treatment-Emergent Adverse Events (Safety) | 10 years
  Evaluated with CTCAE v4.0 or v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Lebbe, MD, PhD, Study Director — AP-HP, Hopital Saint-Louis, centre d'oncodermatologie, Paris; Gaelle Quereux, MD, PhD, Study Director — Nantes University Hospital
Locations (27):
- France (27):
  - CHU d'Amiens, Amiens
  - CH Annecy Genevois, Annecy
  - CHU de Besançon, Besançon
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Avicennes, Bobigny
  - CHU de Bordeaux Hôpital Haut Levêque, Bordeaux
  - CHU de Bordeaux Hôpital Saint-André, Bordeaux
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU de Lille, Lille
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon
  - AP-HM Hopital de la Timone, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice, Nice
  - CHRU de Nîmes, Nîmes
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hopital Saint-Louis, centre d'oncodermatologie, Paris
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Bichat, Paris
  - Assistance Publique - Hôpitaux de Paris (AP-HP), Hôpital Cochin, Paris
  - CHU de Rennes, Rennes
  - CLCC Eugène Marquis, Rennes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plaschka M, Benboubker V, Grimont M, Berthet J, Tonon L, Lopez J, Le-Bouar M, Balme B, Tondeur G, de la Fouchardiere A, Larue L, Puisieux A, Grinberg-Bleyer Y, Bendriss-Vermare N, Dubois B, Caux C, Dalle S, Caramel J. ZEB1 transcription factor promotes immune escape in melanoma. J Immunother Cancer. 2022 Mar;10(3):e003484. doi: 10.1136/jitc-2021-003484. PMID 35288462
- See also: Di Filippo Y. et al., Relevance of body mass index as a predictor of systemic therapy outcomes in metastatic melanoma: analysis of the MelBase French cohort data; Ann Oncol . 2021 Apr;32(4):542-551. doi: 10.1016/j.annonc.2020.12.012. — https://pubmed.ncbi.nlm.nih.gov/33385520/
- See also: Kandel M. et al., Update of survival and cost of metastatic melanoma with new drugs: Estimations from the MelBase cohort ; Eur J Cancer . 2018 Dec;105:33-40. doi: 10.1016/j.ejca.2018.09.026. — https://pubmed.ncbi.nlm.nih.gov/30384014/
- See also: Vallet A. et al., Association of Time From Primary Diagnosis to First Distant Relapse of Metastatic Melanoma With Progression of Disease and Survival ; JAMA Dermatol . 2019 Jun 1;155(6):673-678. doi: 10.1001/jamadermatol.2019.0425. — https://pubmed.ncbi.nlm.nih.gov/31042256/
- See also: Tetu et al.Impact of radiotherapy administered simultaneously with systemic treatment in patients with melanoma brain metastases within MelBase, a French multicentric prospective cohort; Eur J Cancer 2019 May;112:38-46 — https://pubmed.ncbi.nlm.nih.gov/30909072/
- See also: Kandel M et al., Quality-of-life assessment in French patients with metastatic melanoma in real life; Cancer . 2020 Feb 1;126(3):611-618. doi: 10.1002/cncr.32554. — https://pubmed.ncbi.nlm.nih.gov/31639198/
- See also: Huynh S. et al., Combined Therapy with Anti-PD1 and BRAF and/or MEK Inhibitor for Advanced Melanoma: A Multicenter Cohort Study; Cancers (Basel) . 2020 Jun 23;12(6):1666. doi: 10.3390/cancers12061666 — https://pubmed.ncbi.nlm.nih.gov/32585901/
- See also: Carlet C. et al., Late-onset adverse events of anti-PD1 therapy in melanoma patients: An observational study from MELBASE, a nationwide prospective cohort; J Am Acad Dermatol . 2022 Feb;86(2):345-352. doi: 10.1016/j.jaad.2021.06.849 — https://pubmed.ncbi.nlm.nih.gov/34153388/
- See also: Casarotto E. et al., Real-world effectiveness of pembrolizumab in advanced melanoma: analysis of a French national clinicobiological database ; Immunotherapy . 2021 Aug;13(11):905-916. doi: 10.2217/imt-2021-0077 — https://pubmed.ncbi.nlm.nih.gov/34074114/
- See also: Becquart O. et al., Tolerance and Effectiveness of Targeted Therapies in Aged Patients with Metastatic Melanoma ; Cancers (Basel) . 2021 Jun 18;13(12):3042. doi: 10.3390/cancers13123042. — https://pubmed.ncbi.nlm.nih.gov/34207200/
- See also: Girod M. et al., Non-V600E/K BRAF Mutations in Metastatic Melanoma: Molecular Description, Frequency, and Effectiveness of Targeted Therapy in a Large National Cohort ; JCO Precis Oncol . 2022 Nov;6:e2200075. doi: 10.1200/PO.22.00075. — https://pubmed.ncbi.nlm.nih.gov/36356284/
- See also: Placais L. et al.,Risk of irAEs in patients with autoimmune diseases treated by immune checkpoint inhibitors for stage III or IV melanoma: results from a matched case-control study; Ann Rheum Dis 2022 Oct;81(10):1445-1452. doi: 10.1136/ard-2022-222186 — https://pubmed.ncbi.nlm.nih.gov/35788496/
- See also: Rousset P. et al., Impact of systemic therapies in metastatic melanoma of unknown primary: A study from MELBASE, a French multicentric prospective cohort; J Am Acad Dermatol . 2023 Apr;88(4):808-815. doi: 10.1016/j.jaad.2022.11.040 — https://pubmed.ncbi.nlm.nih.gov/36543626/
- See also: Kandel M. et al., Cost-Effectiveness Analysis of Sequential Treatment Strategies for Advanced Melanoma in Real Life in France — https://pubmed.ncbi.nlm.nih.gov/36547139/
- See also: Russo D. et al., Differential gradients of immunotherapy vs targeted therapy efficacy according to the sun-exposure pattern of the site of occurrence of primary melanoma: a multicenter prospective cohort study (MelBase) — https://pubmed.ncbi.nlm.nih.gov/37936607/
- See also: Fournier M. et al., Hyperprogression in advanced melanoma is not restricted to immunotherapy — https://pubmed.ncbi.nlm.nih.gov/37690179/
- See also: Macaire C. et al., Real-life effectiveness on overall survival of continued immune checkpoint inhibition following progression in advanced melanoma: estimation from the Melbase cohort — https://pubmed.ncbi.nlm.nih.gov/39527777/
- See also: Amiot M. et al., When to stop immunotherapy for advanced melanoma: the emulated target trials — https://pubmed.ncbi.nlm.nih.gov/39717261/
- See also: Billard K. et al., The efficacy and safety of first-line metastatic melanoma treatment with ipilimumab + nivolumab versus nivolumab in a real-world setting — https://pubmed.ncbi.nlm.nih.gov/39605282/
- See also: Campo Le Brun I. et al., Methods of nivolumab administration in advanced melanoma: A comparison of patients' clinical outcomes treated with flat dose or weight-adjusted dose, a multicenter observational study — https://pubmed.ncbi.nlm.nih.gov/39645590/